CLINICAL TRIAL: NCT05556525
Title: nCLE Guided Randomized Controlled Trial for Lung Cancer Diagnosis
Brief Title: Needle-Based Confocal Laser Endomicroscopy for Diagnosis of Lung Cancer in Patients With Peripheral Pulmonary Nodules
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: MKT_2021_lung_01; NCI-2022-07660 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21-008276 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2022-09-23; First posted 2022-09-27 (Actual); Results first posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-07

CONDITIONS: Lung Carcinoma
MeSH Terms: conditions — Lung Neoplasms | interventions — Fluorescein

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Raters will be blinded to patient history and cytologic/pathologic diagnosis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm I (EBUS TBNA) (Active Comparator): Patients undergo robotic EBUS TBNA on study.
  Interventions: Procedure: Ultrasound-Guided Transbronchial Needle Aspiration
- Arm II (EBUS TBNA, nCLE, fluorescein) (Experimental): Patients undergo EBUS TBNA, nCLE, and receive fluorescein IV on study.
  Interventions: Other: Fluorescein; Device: Image-Guided Needle Confocal Laser Endomicroscopy; Procedure: Ultrasound-Guided Transbronchial Needle Aspiration

INTERVENTIONS:
Other: Fluorescein — Given IV
  Arms: Arm II (EBUS TBNA, nCLE, fluorescein)
Device: Image-Guided Needle Confocal Laser Endomicroscopy — Undergo nCLE
  Arms: Arm II (EBUS TBNA, nCLE, fluorescein)
Procedure: Ultrasound-Guided Transbronchial Needle Aspiration — Undergo EBUS TBNA
  Other Names: EBUS-TBNA; Endobronchial Ultrasound-Guided Transbronchial Needle Aspiration

SUMMARY:
This clinical trial compares the addition of needle-based confocal laser endomicroscopy (nCLE) and fluorescein to endobronchial ultrasound-guided transbronchial needle aspiration (EBUS TBNA) with EBUS TBNA alone for the diagnosis of lung cancer in patients with peripheral pulmonary nodules. EBUS TBNA is a diagnostic procedure that can be used to sample lung tissue. nCLE is a novel high-resolution imaging technique that uses a laser light to create real-time microscopic images of tissues. It can be integrated into needles allowing real-time cancer detection during endoscopy. Fluorescein is an imaging agent that can be used to visualize tissue. Using nCLE and fluorescein in combination with EBUS TBNA may be more effective in diagnosing lung cancer than using EBUS TBNA alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the first-pass diagnostic yield of the sequential needle passes (rapid on-site evaluation [ROSE]) between the robotic-nCLE-TBNA arm and the robotic-guided arm in peripheral pulmonary nodule (PPNs).

SECONDARY OBJECTIVES:

I. To compare the per-patient diagnostic yield (cumulative pass diagnostic yield: cumulative number of passes until five cumulated passes) of robotic-nCLE-guided TBNA to that of robotic-guided TBNA in PPNs.

II. To compare the proportion of patients with lung cancer treatment in the robotic-nCLE-guided TBNA arm to that of the robotic-guided TBNA arm in PPNs.

III. To compare the proportion of patients with follow-up (video-assisted thoracoscopic surgery [VATS]) or transthoracic needle aspiration (TTNA) or TBNA procedures in the robotic-nCLE-guided TBNA arm to that of the robotic-guided TBNA arm in PPNs.

IV. To compare the number of passes needed to obtain a final diagnosis of robotic-nCLE-guided TBNA to that of robotic-guided TBNA in PPNs.

V. To assess the diagnostic performance (sensitivity, specificity, positive predictive value [PPV], negative predictive value [NPV], accuracy) of the sequential cumulative nCLE passes and the sequential cumulative ROSE passes using the final diagnosis as a reference.

VI. To assess the feasibility by obtaining adequate confocal laser endomicroscopy (CLE) video footage in > 80% of the PPN punctures.

VII. To assess the safety of nCLE imaging, as defined by:

VIIa. The number and frequency of all adverse events (AE)/serious adverse events (SAE) from the start of the procedure until end of 12-month follow-up; VIIb. The number and frequency of nCLE procedure-related AE/SAE from the start of the procedure until end of 12-month follow-up.

VIII. To assess the reproducibility of nCLE criteria to the reference standard. Three nCLE characteristics for the detection of malignancy were identified during Wijmans et al. study:

VIIIa. Dark enlarged pleomorphic cells; VIIIb. Dark cell clusters consist of overlapping cell structures ('dark clumps') and; VIIIc. Continuous movement of the cells in one direction ('directional streaming').

IX. To create an nCLE image atlas for malignant characteristics in PPNs.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo robotic EBUS TBNA on study.

ARM II: Patients undergo EBUS TBNA, nCLE, and receive fluorescein intravenously (IV) on study.

ELIGIBILITY:
Inclusion Criteria:

* >= 21 years of age
* Suspected PPN
* Nodule size in computed tomography (CT) between 8 mm and 30 mm (largest dimension)
* Ability to understand and willingness to sign a written informed consent and Health Insurance Portability and Accountability Act (HIPAA) consent document

Exclusion Criteria:

* Inability or non-willingness to provide informed consent
* Failure to comply with the study protocol
* Patients with known allergy for fluorescein or risk factors for an allergic reaction
* Use of beta-blocker within 24 hours before the start of the bronchoscopic procedure
* Possibly pregnant, pregnant or breastfeeding women
* Patients with hemodynamic instability
* Patients with refractory hypoxemia
* Patients with a therapeutic anticoagulant that cannot be held for an appropriate interval before the procedure
* Patients who are unable to tolerate general anesthesia according to the anesthesiologist
* Patient undergoing chemotherapy
* INTRA-OPERATIVE EXCLUSION/STOPPING CRITERIA:
* The lesions are unable to be localized/confirmed by bronchoscopy
* The procedure will be terminated if the patient develops a significant procedural complication as determined by the treating physician
* The procedure will be terminated if the patient develops hemodynamic instability as determined by the treating physician

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Fernandez-Bussy, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (EBUS TBNA) | Arm II (EBUS TBNA, nCLE, Fluorescein)
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (EBUS TBNA) | Arm II (EBUS TBNA, nCLE, Fluorescein) | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 2 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: First-pass Diagnostic Yield
Description: Calculated as the proportion of patients for which first-pass transbronchial needle aspiration during bronchoscopic procedure yielded a definitive diagnosis out of the total number of patients that have received a diagnostic procedure.
Time Frame: Baseline
Population: The first-pass diagnostic yield could not be determined. Samples obtained at first pass were not separated from remaining samples collected during the procedure, and samples were sent to pathology together, not as per-pass yields. Per-patient (overall) diagnostic yield is reported in outcome 2.
Arm/Group | Arm I (EBUS TBNA) | Arm II (EBUS TBNA, nCLE, Fluorescein)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Per-patient Diagnostic Yield
Description: Calculated as the proportion of patients in whom the bronchoscopic procedure yielded a definitive diagnosis out of the total number of patients that have received a diagnostic procedure. Per patient diagnostic yield of each bronchoscopic procedure will be calculated, and the accuracy of each technique using the final/definitive diagnosis as the reference. The diagnostic yield and accuracy for each method will be compared.
Time Frame: Baseline to 12 months following procedure
Population: For all patients, diagnostic yield was confirmed true during follow-up. The patient who tested negative for malignancy had scar tissue. For the patients who tested positive, one was stable (no change in nodule) during follow-up. The other was diagnosed with adenocarcinoma with enteric origin and metastasis was confirmed; noticed of death was received 10/25/2024 (post follow-up).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (EBUS TBNA) | Arm II (EBUS TBNA, nCLE, Fluorescein)
Number analyzed (Participants) | 2 | 1
Participants
  Negative for carcinoid or malignancy | 0 | 1
  Positive for carcinoid or malignancy | 2 | 0

3. Other Pre Specified Outcome: Clinical Impact of Needle-based Confocal Laser Endomicroscopy (nCLE)
Description: Assessed by determining the proportion of patients with a correct change in definitive diagnosis and the associated change in management plan with nCLE.
Time Frame: Up to 12 months following procedure
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Patients were followed for 12 months (baseline assessment at enrollment to 12-month follow-up assessment/record review). Report of deceased patient was received at 17 months, 1 week (post follow-up).
Arm/Group | Arm I (EBUS TBNA) | Arm II (EBUS TBNA, nCLE, Fluorescein)
All-Cause Mortality (participants affected / at risk) | 1/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 1/2 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (EBUS TBNA) (N=2) | Arm II (EBUS TBNA, nCLE, Fluorescein) (N=1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Non-cardiac Chest Pain (General disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Peripheral Motor Neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Edema Limbs (General disorders) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/25/NCT05556525/Prot_SAP_000.pdf
  • Informed Consent Form (2024-06-21): https://cdn.clinicaltrials.gov/large-docs/25/NCT05556525/ICF_001.pdf